CLINICAL TRIAL: NCT06330727
Title: Effects of Three-Month Coffee Consumption on Metabolic Biomarkers in Adults With Prediabetes and Obesity: a Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Effects of Coffee Consumption on Metabolic Markers in Adults With Prediabetes and Obesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KY20231109-09
Record Dates: First submitted 2024-03-11; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Prediabetes
Keywords: Prediabetes; Obesity; Coffee; Glucose metabolism; Lipid metabolism; Inflammation
MeSH Terms: conditions — Prediabetic State; Obesity; Inflammation | interventions — Coffee; Starch

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coffee capsule (Active Comparator): participants in this arm ingest coffee capsules with 1.8g instant black coffee powder twice daily with breakfast and lunch.
  Interventions: Dietary Supplement: Coffee capsule
- Placebo (Placebo Comparator): participants in this arm consume cornstarch capsules (without coffee) twice daily with breakfast and lunch.
  Interventions: Dietary Supplement: Corn starch capsule

INTERVENTIONS:
Dietary Supplement: Coffee capsule — Take 12 coffee capsules containing 3.6 g instant black coffee powder per day (take 6 coffee capsules twice daily with breakfast and lunch).
  Other Names: 0 sugar 0 fat black coffee, instant black coffee. Product standard code: Q/QC 0001S. Food production license number: SC10644190004159.
  Arms: Coffee capsule
Dietary Supplement: Corn starch capsule — Take 12 placebo capsules containing 3.6 g corn starch per day (take 6 placebo capsules twice daily with breakfast and lunch).
  Other Names: Edible corn starch. Product standard code: GB 31637. Food production license number: SC10313102300041.
  Arms: Placebo

SUMMARY:
Epidemiological studies have shown an inverse association between coffee consumption and risk of type 2 diabetes. However, the randomized controlled trials in prediabetes are limited to evaluate the effects of coffee. The purpose of this study is to investigate the effects of coffee on metabolic factors and inflammation in individuals with prediabetes and obesity. A double-blind, randomized controlled trial is designed to explore the effects of coffee consumption on participants with prediabetes and obesity. A total of 100 eligible participants with prediabetes and obesity will be recruited from the Health Management Center of Nanjing First Hospital. These participants are randomly assigned in a 1:1 ratio to either the coffee capsule group or the control group. The coffee capsule group will be instructed to consume 3.6 g of coffee capsules per day (0.3 g per capsule, 6 capsules per serving, twice a day, once in the morning and once in the middle of the day). The control group will be asked to consume 3.6 g of cornstarch capsules (0.3 g per capsule, 6 capsules per serving, twice a day, once in the morning and once in the middle of the day). 75 g oral glucose tolerance test, 2-week blinded continuous glucose measurement and others will be performed before and after the 3-month intervention. During the three months of intervention, the information on dietary intake, physical activity and sleep of participants will be systematically collected. To comprehensively assess the impact of coffee intake on prediabetes and obesity, we will analyze the effects of coffee capsules on various metabolic and inflammatory markers, including glucose metabolism, lipid profiles, blood pressure, adiponectin, high sensitivity C-reactive protein, interleukin-6, body mass index, body composition, the degree of hepatic steatosis and so on. We will further adjust for potential confounding factors such as lifestyle factors to better understand the underlying biological mechanisms driving this association.

DETAILED DESCRIPTION:
Participants with both prediabetes and obesity who undergo physical examinations at the Health Management Center of Nanjing First Hospital will be recruited for this study. The details of this study design are as follows:

1. Inclusion and exclusion criteria for participants. Inclusion criteria are as follows: 1) Age between 18 and 59 years old; 2) Body mass index (BMI) ≥ 28 kg/m2; 3) No consumption of coffee in the past month; 4) Provide written informed consent; 5) Abnormal glucose tolerance, as per the 1999 WHO diagnostic criteria for prediabetes, includes impaired fasting glucose (IFG), impaired glucose tolerance (IGT) or a combination of both, with blood glucose fluctuations within an abnormal range (fasting blood glucose ≥6.1 mmol/L but <7.0 mmol/L, and/or 2-hour glucose tolerance blood glucose ≥7.8 mmol/L but <11.1 mmol/L). The exclusion criteria for participants include individuals who 1) have been diagnosed with diabetes or are taking anti-diabetic drugs; 2) have a history of diseases such as cancer, liver and kidney dysfunction, existing cardiovascular and cerebrovascular diseases, and other diseases that may affect glucose and lipid metabolism; 3) self-report gastrointestinal reaction or intolerance to coffee and reject coffee consumption; 4) are pregnant or planning to become pregnant in the near future; 5) are deemed unsuitable to participate in this study by researcher believes that they are not to participate in this study.

2. Sample size calculation: Based on the estimation of research purpose, research design, expected effect size, and statistical analysis method, the sample size is determined to be 100 cases, including fifty cases in the intervention group and fifty cases in the control group.

3. Definition of the intervention group and placebo group: the intervention group serves as the coffee capsule group, and will receive 3.6 g of coffee capsules per day (0.3 g/capsule, 6 capsules/time, 2 times/day, once in the morning and once in the middle of the day). The placebo group (control group) is required to consume 3.6 g of cornstarch capsules per day (0.3 g/capsule, 6 capsules/time, 2 times/day, once in the morning and once in the middle of the day).

4. Follow-up and data collection: this follow-up period will span three months. Before and after the 3-month intervention the participants will partake in:

1. regular assessments. Demographic characteristics and medical information will be collected, including age, gender, occupation, education level, income, medication history (hormones, contraceptives, etc.), and family history of chronic diseases. Besides, using questionnaires, we also collect lifestyle information such as smoking, drinking, diet intake, physical activity, and sleep of participants. Specifically, the Simplified Food Frequency Questionnaire (FFQ25) and 24-hour Diet Record Questionnaire (DR) are employed to assess the dietary intake of participants in the past six months and the previous 24 hours (one day each in the middle of the week and on the weekend), respectively. International Physical Activity Questionnaire (IPAQ) is utilized to assess various aspects of physical activity, including time, frequency, and intensity. The sleep information (sleep time, sleep quality, etc.) is evaluated by Pittsburgh sleep quality index (PSQI).
2. A 75 g oral glucose tolerance test (75 g-OGTT). Blood samples are taken fasting and 30, 120 minutes after the glucose load. Blood samples are analyzed for glucose, insulin, C-peptide, and glucagon.
3. 2-week continuous glucose measurement using blinded continuous glucose monitor/sensor on upper arm.
4. Fasting blood samples: glycated hemoglobin (HbA1c), total cholesterol, high-density lipoprotein-cholesterol (HDL-C), low-density lipoprotein-cholesterol (LDL-C), triglycerides, high sensitivity C-reactive protein (CRP), interleukin 6 (IL-6).
5. Furthermore, blood pressure, transient hepatic elastography for the assessment of fatty liver degree, body composition analysis, and heart rhythm variation analysis are collected using corresponding instrument and equipment inspection. Additionally, blood, urine, and stool samples will be collected for further analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 59 years old;
2. Diagnosis of Prediabetes according to the WHO criteria (fasting glucose=6.1-6.9 mmol/L and/or 2-hour post-OGTT glucose=7.8- 11.0 mmol/L);
3. Body mass index ( BMI ) ≥ 28kg/m2;
4. No coffee intake in the past month;
5. Provide written informed consent and be willing to participate.

Exclusion Criteria:

1. Patients with diagnosis of diabetes, or taking anti-diabetic medication;
2. Patients with cardiovascular or cerebrovascular diseases, cancer, renal disease, liver disease, other chronic diseases affecting glucose and lipid metabolism, etc;
3. Participants with known hypersensitivity or intolerance to coffee, or unwilling to accept coffee;
4. Pregnancy, planned pregnancy, or lactation;
5. Investigators, for any reason, consider the participants inappropriate for the study (e.g., uncontrolled bipolar disease).

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Continuous glucose monitoring parameters | at baseline, after three-month intervention
  14 days blinded intermittent-scanned continuous glucose monitoring (CGM): the FreeStyle Libre Pro system is utilized to record glycemic data, with the readout of the device exclusively performed by researchers. During the day, participants will be blinded to their glucose values.
glucose from a 75 g-oral glucose tolerance test （mmol/L） | at baseline, after one-month intervention, after three-month intervention
  Blood samples will be drawn at time points 0 min, 30 min, 120 min for glucose measurements during a 75 g-oral glucose tolerance test (75 g-OGTT).
  Incremental glucose area under the curve (gAUC) will be calculated using the trapezoidal method.
insulin from a 75 g-oral glucose tolerance test （pmol/L） | at baseline, after one-month intervention, after three-month intervention
  Blood samples will be drawn at time points 0 min, 30 min, 120 min for insulin measurements during a 75 g-oral glucose tolerance test (75 g-OGTT).
  Incremental insulin area under the curve (iAUC) will be calculated using the trapezoidal method.
C-peptide from a 75 g-oral glucose tolerance test (ng/ml) | at baseline, after one-month intervention, after three-month intervention
  Blood samples will be drawn at time points 0 min, 30 min, 120 min for C-peptide measurements during a 75 g-oral glucose tolerance test (75 g-OGTT).
glucagon from a 75 g-oral glucose tolerance test（pmol/L） | at baseline, after one-month intervention, after three-month intervention
  Blood samples will be drawn at time points 0 min, 30 min, 120 min for glucagon measurements during a 75 g-oral glucose tolerance test (75 g-OGTT).
Glycated hemoglobin (HbA1c) ( % ) | at baseline, after three-month intervention
  Reflect the levels of blood sugar in the past two to three months.
Fasting total cholesterol (mmol/L) | at baseline, after one-month intervention, after three-month intervention
  Serum total cholesterol concentrations under fasting conditions.
Fasting high-density lipoprotein-cholesterol (mmol/L) | at baseline, after one-month intervention, after three-month intervention
  Serum high-density lipoprotein-cholesterol (HDL-C) concentrations under fasting conditions.
Fasting low-density lipoprotein-cholesterol (mmol/L) | at baseline, after one-month intervention, after three-month intervention
  Serum low-density lipoprotein-cholesterol ( LDL-C) concentrations under fasting conditions.
Fasting triglycerides (mmol/L) | at baseline, after one-month intervention, after three-month intervention
  Serum triglycerides concentrations under fasting conditions.

SECONDARY OUTCOMES:
C-reactive protein | at baseline, after one-month intervention, after three-month intervention
  Serum levels of inflammatory factors: high-sensitivity C-reactive protein (CRP).
Interleukin-6 | at baseline, after one-month intervention, after three-month intervention
  Serum levels of inflammatory factors: interleukin-6 (IL-6).
Body mass index ( kg/m^2) | at baseline, after one-month intervention, after three-month intervention
  Calculation of body mass index (BMI) using body weight and height.
Fat mass (FM) | at baseline, after one-month intervention, after three-month intervention
  Assessed using an InBody bioelectrical impedance analyzer.
body fat percentage (BF) | at baseline, after one-month intervention, after three-month intervention
  Assessed using an InBody bioelectrical impedance analyzer.
visceral fat | at baseline, after one-month intervention, after three-month intervention
  Assessed using an InBody bioelectrical impedance analyzer.
skeletal muscle mass (SMM) | at baseline, after one-month intervention, after three-month intervention
  Assessed using an InBody bioelectrical impedance analyzer.
fat-free mass (FFM) | at baseline, after one-month intervention, after three-month intervention
  Assessed using an InBody bioelectrical impedance analyzer.
Adiponectin | at baseline, after one-month intervention, after three-month intervention
  high-molecular-weight adiponectin
Systolic blood pressure（mmHg） | at baseline, after one-month intervention, after three-month intervention
  After 20 min of rest, blood pressure will be measured between 8:00 and 9:00 in the morning by an experienced nurse and the average of three consecutive measurements will be recorded.
Diastolic blood pressure（mmHg） | at baseline, after one-month intervention, after three-month intervention
  After 20 min of rest, blood pressure will be measured between 8:00 and 9:00 in the morning by an experienced nurse and the average of three consecutive measurements will be recorded.
Heart rate （bpm） | at baseline, after one-month intervention, after three-month intervention
  After 20 min of rest, heart rate will be measured between 8:00 and 9:00 in the morning by an experienced nurse and the average of three consecutive measurements will be recorded.
Controlled attenuation parameter (CAP) | at baseline, after one-month intervention, after three-month intervention
  Controlled attenuation parameter (CAP) by transient hepatic elastography (THE) assesses the degree of hepatic steatosis.
Standard deviation of heart rate variability (SDNN) | at baseline, after one-month intervention, after three-month intervention
  Heart Rhythm Variation Analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Wang, M.D.,phD., Principal Investigator — Health Management Center of Nanjing First Hospital
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ding M, Bhupathiraju SN, Chen M, van Dam RM, Hu FB. Caffeinated and decaffeinated coffee consumption and risk of type 2 diabetes: a systematic review and a dose-response meta-analysis. Diabetes Care. 2014 Feb;37(2):569-86. doi: 10.2337/dc13-1203. PMID 24459154
- [Background] Scheen AJ, Letiexhe MR, Ernest P. [Prevention of type 2 diabetes: lifestyle changes or pharmacological interventions?]. Rev Med Liege. 2003 Apr;58(4):206-10. French. PMID 12868322
- [Background] Schulze MB, Hu FB. Primary prevention of diabetes: what can be done and how much can be prevented? Annu Rev Public Health. 2005;26:445-67. doi: 10.1146/annurev.publhealth.26.021304.144532. PMID 15760297
- [Background] Magis D, Geronooz I, Scheen AJ. [Smoking, insulin resistance and type 2 diabetes]. Rev Med Liege. 2002 Sep;57(9):575-81. French. PMID 12440345
- [Background] Higdon JV, Frei B. Coffee and health: a review of recent human research. Crit Rev Food Sci Nutr. 2006;46(2):101-23. doi: 10.1080/10408390500400009. PMID 16507475
- [Background] van Dam RM. Coffee and type 2 diabetes: from beans to beta-cells. Nutr Metab Cardiovasc Dis. 2006 Jan;16(1):69-77. doi: 10.1016/j.numecd.2005.10.003. Epub 2005 Dec 13. PMID 16399494
- [Background] Bellou V, Belbasis L, Tzoulaki I, Evangelou E. Risk factors for type 2 diabetes mellitus: An exposure-wide umbrella review of meta-analyses. PLoS One. 2018 Mar 20;13(3):e0194127. doi: 10.1371/journal.pone.0194127. eCollection 2018. PMID 29558518
- [Background] Kondo Y, Goto A, Noma H, Iso H, Hayashi K, Noda M. Effects of Coffee and Tea Consumption on Glucose Metabolism: A Systematic Review and Network Meta-Analysis. Nutrients. 2018 Dec 27;11(1):48. doi: 10.3390/nu11010048. PMID 30591664
- [Background] Bae JM. Coffee consumption and risk of type 2 diabetes mellitus in Asians: A meta-epidemiological study of population-based cohort studies. World J Diabetes. 2021 Jun 15;12(6):908-915. doi: 10.4239/wjd.v12.i6.908. PMID 34168737
- [Background] Di Maso M, Boffetta P, Negri E, La Vecchia C, Bravi F. Caffeinated Coffee Consumption and Health Outcomes in the US Population: A Dose-Response Meta-Analysis and Estimation of Disease Cases and Deaths Avoided. Adv Nutr. 2021 Jul 30;12(4):1160-1176. doi: 10.1093/advances/nmaa177. PMID 33570108
- [Background] Osama H, Abdelrahman MA, Madney YM, Harb HS, Saeed H, Abdelrahim MEA. Coffee and type 2 diabetes risk: Is the association mediated by adiponectin, leptin, c-reactive protein or Interleukin-6? A systematic review and meta-analysis. Int J Clin Pract. 2021 Jun;75(6):e13983. doi: 10.1111/ijcp.13983. Epub 2021 Jan 21. PMID 33400346
- [Background] Shahinfar H, Jayedi A, Khan TA, Shab-Bidar S. Coffee consumption and cardiovascular diseases and mortality in patients with type 2 diabetes: A systematic review and dose-response meta-analysis of cohort studies. Nutr Metab Cardiovasc Dis. 2021 Aug 26;31(9):2526-2538. doi: 10.1016/j.numecd.2021.05.014. Epub 2021 May 24. PMID 34112583
- [Background] Carlstrom M, Larsson SC. Coffee consumption and reduced risk of developing type 2 diabetes: a systematic review with meta-analysis. Nutr Rev. 2018 Jun 1;76(6):395-417. doi: 10.1093/nutrit/nuy014. PMID 29590460
- [Background] Bhupathiraju SN, Pan A, Manson JE, Willett WC, van Dam RM, Hu FB. Changes in coffee intake and subsequent risk of type 2 diabetes: three large cohorts of US men and women. Diabetologia. 2014 Jul;57(7):1346-54. doi: 10.1007/s00125-014-3235-7. Epub 2014 Apr 26. PMID 24771089
- [Background] van Dam RM, Feskens EJ. Coffee consumption and risk of type 2 diabetes mellitus. Lancet. 2002 Nov 9;360(9344):1477-8. doi: 10.1016/S0140-6736(02)11436-X. PMID 12433517
- [Background] Bidel S, Silventoinen K, Hu G, Lee DH, Kaprio J, Tuomilehto J. Coffee consumption, serum gamma-glutamyltransferase and risk of type II diabetes. Eur J Clin Nutr. 2008 Feb;62(2):178-85. doi: 10.1038/sj.ejcn.1602712. Epub 2007 Mar 7. PMID 17342160
- [Background] Greenberg JA, Boozer CN, Geliebter A. Coffee, diabetes, and weight control. Am J Clin Nutr. 2006 Oct;84(4):682-93. doi: 10.1093/ajcn/84.4.682. PMID 17023692
- [Background] Doo T, Morimoto Y, Steinbrecher A, Kolonel LN, Maskarinec G. Coffee intake and risk of type 2 diabetes: the Multiethnic Cohort. Public Health Nutr. 2014 Jun;17(6):1328-36. doi: 10.1017/S1368980013000487. Epub 2013 Feb 27. PMID 23442347
- [Background] Greenberg JA, Axen KV, Schnoll R, Boozer CN. Coffee, tea and diabetes: the role of weight loss and caffeine. Int J Obes (Lond). 2005 Sep;29(9):1121-9. doi: 10.1038/sj.ijo.0802999. PMID 15925959
- [Background] Iso H, Date C, Wakai K, Fukui M, Tamakoshi A; JACC Study Group. The relationship between green tea and total caffeine intake and risk for self-reported type 2 diabetes among Japanese adults. Ann Intern Med. 2006 Apr 18;144(8):554-62. doi: 10.7326/0003-4819-144-8-200604180-00005. PMID 16618952
- [Background] Karabegovic I, Portilla-Fernandez E, Li Y, Ma J, Maas SCE, Sun D, Hu EA, Kuhnel B, Zhang Y, Ambatipudi S, Fiorito G, Huang J, Castillo-Fernandez JE, Wiggins KL, de Klein N, Grioni S, Swenson BR, Polidoro S, Treur JL, Cuenin C, Tsai PC, Costeira R, Chajes V, Braun K, Verweij N, Kretschmer A, Franke L, van Meurs JBJ, Uitterlinden AG, de Knegt RJ, Ikram MA, Dehghan A, Peters A, Schottker B, Gharib SA, Sotoodehnia N, Bell JT, Elliott P, Vineis P, Relton C, Herceg Z, Brenner H, Waldenberger M, Rebholz CM, Voortman T, Pan Q, Fornage M, Levy D, Kayser M, Ghanbari M. Epigenome-wide association meta-analysis of DNA methylation with coffee and tea consumption. Nat Commun. 2021 May 14;12(1):2830. doi: 10.1038/s41467-021-22752-6. PMID 33990564
- [Background] Hang D, Kvaerner AS, Ma W, Hu Y, Tabung FK, Nan H, Hu Z, Shen H, Mucci LA, Chan AT, Giovannucci EL, Song M. Coffee consumption and plasma biomarkers of metabolic and inflammatory pathways in US health professionals. Am J Clin Nutr. 2019 Mar 1;109(3):635-647. doi: 10.1093/ajcn/nqy295. PMID 30834441
- [Background] Shang F, Li X, Jiang X. Coffee consumption and risk of the metabolic syndrome: A meta-analysis. Diabetes Metab. 2016 Apr;42(2):80-7. doi: 10.1016/j.diabet.2015.09.001. Epub 2015 Oct 1. PMID 26431818
- [Background] Poole R, Kennedy OJ, Roderick P, Fallowfield JA, Hayes PC, Parkes J. Coffee consumption and health: umbrella review of meta-analyses of multiple health outcomes. BMJ. 2017 Nov 22;359:j5024. doi: 10.1136/bmj.j5024. PMID 29167102
- [Background] Grosso G, Godos J, Galvano F, Giovannucci EL. Coffee, Caffeine, and Health Outcomes: An Umbrella Review. Annu Rev Nutr. 2017 Aug 21;37:131-156. doi: 10.1146/annurev-nutr-071816-064941. PMID 28826374
- [Background] Pan MH, Tung YC, Yang G, Li S, Ho CT. Molecular mechanisms of the anti-obesity effect of bioactive compounds in tea and coffee. Food Funct. 2016 Nov 9;7(11):4481-4491. doi: 10.1039/c6fo01168c. PMID 27722362
- [Background] Martini D, Del Bo' C, Tassotti M, Riso P, Del Rio D, Brighenti F, Porrini M. Coffee Consumption and Oxidative Stress: A Review of Human Intervention Studies. Molecules. 2016 Jul 28;21(8):979. doi: 10.3390/molecules21080979. PMID 27483219
- [Background] Shi X, Xue W, Liang S, Zhao J, Zhang X. Acute caffeine ingestion reduces insulin sensitivity in healthy subjects: a systematic review and meta-analysis. Nutr J. 2016 Dec 28;15(1):103. doi: 10.1186/s12937-016-0220-7. PMID 28031026
- [Background] Ding M, Satija A, Bhupathiraju SN, Hu Y, Sun Q, Han J, Lopez-Garcia E, Willett W, van Dam RM, Hu FB. Association of Coffee Consumption With Total and Cause-Specific Mortality in 3 Large Prospective Cohorts. Circulation. 2015 Dec 15;132(24):2305-15. doi: 10.1161/CIRCULATIONAHA.115.017341. Epub 2015 Nov 16. PMID 26572796